CLINICAL TRIAL: NCT06655740
Title: A Pilot Human Study of the Safety, Tolerability and Effectiveness of the Aqua Medical Circumferential RF Vapor (RFV) Ablation System for Duodenal Mucosal Ablation for the Management of Insulin Requiring Type-2 Diabetes Mellitus
Brief Title: Safety, Tolerability, and Effectiveness of Duodenal Mucosal RF Vapor Ablation for Insulin Elimination in Type-2 Diabetes
Acronym: STEAM-IE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-1022-SA
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study arm- RF Vapor Ablation arm (Experimental): This is a single arm study. All enrolled patients will be included in this arm
  Interventions: Device: RF Vapor Ablation

INTERVENTIONS:
Device: RF Vapor Ablation — RF Vapor ablation of the duodenum

SUMMARY:
The purpose of this study is to determine whether RFVA of the duodenal mucosa with or without the combination of Semaglutide is a safe and effective treatment to remove the need for insulin therapy among patients with T2D who are on stable doses of insulin.

DETAILED DESCRIPTION:
This is a prospective, open-label pilot, to determine safety and efficacy of step-up therapy with RFVA and Semaglutide

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old but ≤ 65 years old. (Women of childbearing potential must be using one acceptable methods of contraception throughout the study.)
2. Diagnosed with type 2 diabetes mellitus for ≥1 year but ≤ 8 years duration.
3. Glycated haemoglobin ≤ 8.0% (64 mmol/mol).
4. Fasting serum C-peptide ≥ 0.6 ng/mL.
5. Body mass index ≥ 27.5 and ≤ 42.5 kg/m2.
6. On a daily insulin (basal or combined with short-acting) for at least three months, with a dose ≤ 0.6 U/kg, with a stable dose (≤ 20%) over the last month.
7. Able to comply with study requirements and understand and sign the informed consent form.

Exclusion Criteria:

1. Diagnosis of Type 1 diabetes mellitus
2. Any history of diabetic ketoacidosis or hyperosmolar nonketotic coma
3. Current use of insulin pump.
4. Current, or within the last 3 months, use of a GLP-1 analogue.
5. Current use of a long-acting sulphonylureas (e.g. glibenclamide, chlorpropamide, glimepiride, glyburide)
6. History of severe hypoglycemia (more than 1 severe hypoglycemic event, as defined by need for third-party assistance, in the last year).
7. Known autoimmune disease, including but not limited to celiac disease, duodenal Crohn disease or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other systemic autoimmune connective tissue disorder.
8. Previous gastrointestinal surgery that could limit treatment of the duodenum such as Billroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions. (Prior laparoscopic sleeve gastrectomy (LSG) will not be an exclusion).
9. History of pancreatitis (acute or chronic).
10. Known diabetic gastroparesis.
11. Persistent anaemia, defined as haemoglobin ≤ 9 g/dL
12. Known active hepatitis or active liver disease.
13. Acute gastrointestinal illness in the previous 7 days.
14. Known history of severe irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease.
15. Known history of a structural or functional disorder of the esophagus that may impede passage of the device through the gastrointestinal tract or increase risk of esophageal damage during an endoscopic procedure, including moderate-severe (Grade C or D) esophagitis, dysphagia due to achalasia or stricture/stenosis, esophageal varices, esophageal perforation, or any other disorder of the esophagus.
16. Upper gastrointestinal conditions such as active ulcers, polyps, varices, strictures, congenital or acquired duodenal telangiectasia.
17. Current use of anticoagulation therapy (e.g. warfarin) or direct-acting oral anticoagulants (e.g. rivaroxaban, apixaban, edoxaban and dabigatran) that cannot be discontinued for 3-5 days before and 7 days after the procedure.
18. Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 5 days before and 7 days after the procedure.
19. Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of acetaminophen and low dose aspirin is allowed.
20. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the baseline visit.
21. Use of drugs known to affect gastrointestinal motility (e.g. Metoclopramide)
22. Use of weight loss medications such as Sibutramine (e.g. Meridia), Orlistat (e.g. Xenical), Phentermine or over-the-counter weight loss medications (prescription medication)
23. Significant cardiovascular disease, including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within 6 months prior to the Screening Visit.
24. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
25. Uncontrolled thyroid disease
26. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic).
27. Estimated glomerular filtration rate (eGFR) ≤ 45 ml/min/1.73m2 (estimated by MDRD).
28. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the participant a poor candidate for clinical trial participation in the opinion of the investigator.
29. Active illicit substance abuse or alcoholism (>2 drinks/day regularly)
30. Active malignancy within the last 5 years (excluding non-melanoma skin cancers)
31. Active systemic infection
32. Women who are currently breastfeeding.
33. Pregnancy or wish to get pregnant in the next year.
34. Participating in another ongoing clinical trial of an investigational drug or device.
35. Any other mental or physical condition which, in the opinion of the study investigator, makes the participant a poor candidate for clinical trial participation.
36. Critically ill or has a life expectancy < 3 years.
37. Use of heart pacemaker or other electronic device implants
38. General contraindications to deep or conscious sedation, general anesthesia, high risk as determined by anesthesiologist (e.g., ASA score 4 or higher), or contraindications to upper GI endoscopy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | 1 month
  Number of subjects with reported device or procedure related SAEs or UADEs.
Efficacy Endpoint | 168 days
  Percentage of patients free of insulin at 168 days post RF vapor ablation with an HbA1c ≤ 7.5% (58 mmol/mol)

SECONDARY OUTCOMES:
Technical success of duodenal mucosal ablation using RFVA | 1 month
  The percentage of patients who underwent the procedure and received therapy to ≥ 6cm.
Procedure time | 1 month
  Procedure time of duodenal mucosal ablation, defined as the interval between catheter insertion and removal following completion of the procedure.
Proportion of patients who remain free of insulin and Semaglutide | 24 weeks
  - Proportion of patients who remain free of insulin and Semaglutide at 168 days (24 weeks) following RFVA with a HbA1c ≤ 7.5% (58 mmol/mol)
Absolute change in HbA1c | 84 days
  Absolute change in HbA1c at 84 days post-procedure.
Absolute change in HbA1c by visit over time | 168 days
  Absolute change in HbA1c by visit over time
Change in fasting plasma glucose from baseline | 168 days
  Change in fasting plasma glucose from baseline to 84 and 168 days post-procedure.
Change in fasting plasma glucose by visit over time | 168 days
  Change in fasting plasma glucose by visit over time (up to 168 days post-procedure).
Change in HOMA-IR by visit over time | 168 days
  Change in HOMA-IR by visit over time (up to 168 days post- procedure).
Change in alanine transaminase | 168 days
  Change in alanine transaminase from baseline to 168 days post-procedure.
Change in aspartate transaminase | 168 days
  Change in aspartate transaminase from baseline to 168 days post-procedure.
Change in fibrosis index 4 (FIB-4) score | 168 days
  Change in fibrosis index 4 (FIB-4) score between baseline to 84, baseline to 168 days and 84 to 168 days post-procedure.
Change in non-alcoholic fatty liver disease (NAFLD) fibrosis score | 168 days
  Change in non-alcoholic fatty liver disease (NAFLD) fibrosis score between baseline to 84, baseline to 168 days and 84 to 168 days post-procedure.
Change in BMI | 168 days
  Change in body mass index (BMI) between baseline to 84 and 168 days post-procedure.
Reduction in insulin dose from baseline | 168 days
  Reduction in mean and median dose of insulin from baseline to 168 days post procedure.
Proportion of subjects with ≥50% reduction in their insulin dose at 168 days | 168 days
  Proportion of subjects with ≥50% reduction in their insulin dose at 168 days post- procedure.
Percentage of patients who remain off insulin | 168 days
  Percentage of patients who remain off insulin at 168 days post-procedure.
Proportion of patients who can tolerate semaglutide without need for discontinuation | 168 days
  Proportion of patients who can tolerate semaglutide without need for discontinuation up to 168 days post-procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Colonial, Santiago, Chile